CLINICAL TRIAL: NCT00243841
Title: Multi-institution Phase I/II Dose Escalation Study of Hypofractionated Stereotactic Body Radiation Therapy for Primary Hepatocellular Carcinoma
Brief Title: Dose Escalation Study for Primary Hepatocellular Carcinoma
Acronym: SBF-HCC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Indiana University School of Medicine (Other)
Collaborators: University of Colorado, Denver (Other)
Responsible Party: Principal Investigator, Mark Langer, Professor of Clinical Radiation Oncology, Indiana University School of Medicine
Organization: Indiana University (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0404-20 (1011003002)
Record Dates: First submitted 2005-10-21; First posted 2005-10-25 (Estimated); Results first posted 2018-12-13 (Actual); Last update posted 2018-12-13 (Actual); Status verified 2018-11

CONDITIONS: Carcinoma, Hepatocellular
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — Radiosurgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Radiation Treatment Arm :A (Experimental): Patients with a score of Childs A Will receive 3 fractions of radiation over 5-10 days
  Interventions: Radiation: Stereotactic Body Radiation
- Radiation Treatment Arm: B (Experimental): Patients with a score of Childs B will receive 5 fractions of radiation over 2-6 weeks.
  Interventions: Radiation: Stereotactic Body Radiation

INTERVENTIONS:
Radiation: Stereotactic Body Radiation — Arm A: Childs A - receive 3 fractions. Arm B: Childs B - receive 5 fractions.
  Other Names: Stereotactic Body Radiation Treatments

SUMMARY:
The purpose of this study is to determine the maximum tolerated dose of limited fractions of large dose radiation in an effort to achieve a biologically potent cancer therapy in selected patients with primary hepatocellular carcinoma.

DETAILED DESCRIPTION:
Despite recent advances in early detection and diagnosis, only 30-40% of patients with hepatocellular carcinoma may benefit from radical therapies. Liver transplantation offers the best chance for cure. Surgical resection has been the only other potentially curative option, but the majority of patients are not candidates for resection. This reflects the usual comorbidity of severe underlying liver disease that either precludes surgery or makes the surgical approach extremely dangerous.

ELIGIBILITY:
Inclusion Criteria:

Evaluation by the Surgery and/or Liver Transplant Team has been performed and the patient is not considered a candidate for either "standard" therapy to target area (upper abdomen)

* Adequate liver function defined as:

  * total bilirubin < 3mg/dl, albumin > 2.5 g/dl
  * normal PT/PTT unless on anticoagulants
  * mild elevation of liver enzymes acceptable (must be less than three times upper limit of normal)
* Adequate renal function (creatinine < 1.8 mg/dl or creatinine clearance ≥ 50 ml/min)
* Adequate bone marrow reserve:

  * ANC count ≥ 1500 mm3
  * Platelets ≥ 50,000/mm3
  * Hemoglobin > 9 g/dL

NOTE: Lab values must be obtained within 2 weeks prior to being registered for protocol therapy.

Exclusion Criteria:

* No history of systemic lupus erythematous, rheumatoid arthritis, systemic sclerosis or scleroderma
* No chemotherapy within 14 days before radiotherapy (chemotherapy may cause transient hepatitis with hepatomegaly)
* No subsequent chemotherapy planned within 2 weeks of radiotherapy
* No active liver infection
* No acute Hepatitis. Definition of active disease:

  * Hepatitis A: Acute hepatitis determined by presence of Anti-HAV- IgM
  * Hepatitis B:

    1. HBsAg (HB surface Antigen): present in patients with acute and chronic hepatitis
    2. HBV DNA present in patients with active viral replication in amounts greater than 100,000 copies
    3. HBeAg is present in wild type HBV infection and suggests active replication
    4. Anti-HBs: Antibody against HBsAg appears after HBV infections and confers immunity
    5. Anti-HBc-IgM: Antibody against HBcAg, fraction IgM, present in acute infection and often could be detected during periods of high viral replication in chronic disease
    6. Anti-HBc-IgG: is present in chronic disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 77 (Actual)
Dates: Start 2004-05; Primary Completion 2016-12-31 (Actual); Study Completion 2016-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark Langer, MD, Principal Investigator — Indiana University School of Medicine
Locations (1):
- Indiana University Department of Radiation Oncology, Indianapolis, Indiana, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: This is a Phase I/II study. Phase I is a dose finding study, and Phase II will use the doses determined by the Phase I portion to further look at efficacy. During Phase I, it was determined to look at Childs A patients separately from Childs B patients. Patients who were Childs B required a dose reduction during Phase I.
Groups:
- Phase I: 36 Gy: Patients will receive 1200 cGy x 3 fractions of radiation
- Phase I: 42 Gy: Patients will receive 1400 cGy x 3 fractions of radiation
- Phase I: 40 Gy: Patients will receive 800 cGy x 5 fractions of radiation for Childs B only (dose reduction)
- Phase I: 48 Gy: Patients will receive 1600 cGy x 3 fractions of radiation for Childs A only
- Phase II Childs A: Patients in Phase II with a score of Childs A Will receive 3 fractions (48 Gy) of radiation over 5-10 days
- Phase II Childs B: Patients in Phase II with a score of Childs B will receive 5 fractions (40 Gy) of radiation over 2-6 weeks.
Period: Overall Study
Arm/Group | Phase I: 36 Gy | Phase I: 42 Gy | Phase I: 40 Gy | Phase I: 48 Gy | Phase II Childs A | Phase II Childs B
Started | 3 | 6 | 5 | 3 | 39 | 21
Completed | 3 | 6 | 4 | 3 | 39 | 19
Not Completed | 0 | 0 | 1 | 0 | 0 | 2
Not completed — Physician Decision | 0 | 0 | 1 | 0 | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Phase I: Dose escalation to 48 Gy (16Gy/fraction) in Childs A and to 42 Gy (14 Gy/fraction) down to 40 Gy (8Gy/fraction) for Childs B
- Total: Total of all reporting groups
Arm/Group | Phase I | Phase II Childs A | Phase II Childs B | Total
Number analyzed (Participants) | 17 | 39 | 21 | 77
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 10 | 27 | 17 | 54
  >=65 years | 7 | 12 | 4 | 23
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.8 (9.76) | 60.9 (10.62) | 58.5 (7.55) | 60.2 (9.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 11 | 4 | 16
  Male | 16 | 28 | 17 | 61
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 1 | 1
  Not Hispanic or Latino | 16 | 38 | 20 | 74
  Unknown or Not Reported | 1 | 1 | 0 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 2 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 2 | 7 | 2 | 11
  White | 15 | 30 | 19 | 64
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients With DLTs
Description: Number of patients experiencing a Dose Limiting Toxicity during the Phase I portion of the trial.
Time Frame: 6 weeks
Population: All patients who received treatment in Phase I
Measure: Count of Participants; unit: Participants
Arm/Group | Phase I: 36 Gy | Phase I: 42 Gy | Phase I: 40 Gy | Phase I: 48 Gy
Number analyzed (Participants) | 3 | 6 | 5 | 3
Participants | 0 | 2 | 1 | 0

2. Primary Outcome: 6 Month Local In-field Control
Description: Percent of patients and the 95% Binomial Confidence interval who were free of in-field progression at 6 months following treatment for the patients in Phase II
Time Frame: 6 months
Population: All patients who received treatment and had a post-baseline assessment.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Phase II Childs A | Phase II Childs B
Number analyzed (Participants) | 39 | 21
percentage of participants | 92.3 [79.1 to 98.4] | 87.5 [61.7 to 98.5]

3. Secondary Outcome: Time to In-field Failure
Description: Kaplan-Meier Analyses will be used to calculate the median and 95% Confidence Interval for the time until in-field failure. This will be calculated from the time of treatment until the time of in-field failure. If a patient did not have in-field failure, the patient will be censored at their last evaluation date.
Time Frame: up to 4 yrs
Population: All pts who received treatment and had a post-baseline assessment
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Phase II Childs A | Phase II Childs B
Number analyzed (Participants) | 39 | 19
months | NA [NA to NA] — insufficient number of participants with events to estimate | 32.2 [32.2 to NA] — insufficient number of participants with events to estimate

4. Secondary Outcome: Overall Survival
Description: Kaplan-Meier Analysis will be used to calculate the median and 95% CI for overall survival. This will be calculated from the time of treatment until death. If a patient did not die, the patient will be censored at their last known alive date.
Time Frame: Up to 8 years
Population: all patients who received treatment and had a post-baseline assessment
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Radiation Treatment Arm :A | Radiation Treatment Arm: B
Number analyzed (Participants) | 39 | 19
months | 50.43 [30.88 to 68.59] | 21.40 [10.45 to NA] — insufficient number of participants with events to estimate

5. Secondary Outcome: Phase II: Number of Patients With Treatment Related Grade 3 or 4 Adverse Events
Description: Number of unique patients who had grade 3 or 4 adverse events that were possibly, probably or definitely related to study treatment.
Time Frame: up to 4 years
Population: All patients who received treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Phase II Childs A | Phase II Childs B
Number analyzed (Participants) | 39 | 21
Participants | 5 | 9

ADVERSE EVENTS:
Time Frame: up to 4 years
Arm/Group | Phase I: 36 Gy | Phase I: 42 Gy | Phase I: 40 Gy | Phase I: 48 Gy | Phase II Childs A | Phase II Childs B
All-Cause Mortality (participants affected / at risk) | 3/3 | 4/6 | 4/5 | 2/3 | 19/39 | 13/21
Serious Adverse Events (participants affected / at risk) | 1/3 | 1/6 | 1/5 | 1/3 | 1/39 | 1/21
Other Adverse Events (participants affected / at risk) | 3/3 | 6/6 | 5/5 | 3/3 | 39/39 | 21/21
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Phase I: 36 Gy (N=3) | Phase I: 42 Gy (N=6) | Phase I: 40 Gy (N=5) | Phase I: 48 Gy (N=3) | Phase II Childs A (N=39) | Phase II Childs B (N=21)
Hemoglobin (Investigations) | 0 | 0 | 1 | 0 | 1 | 0
potassium (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1
Leukocytes (total WBC) (Investigations) | 0 | 0 | 0 | 1 | 0 | 0
Platelets (Investigations) | 0 | 0 | 1 | 1 | 0 | 0
Cardiac arhythmia - other (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0
Gastrointestinal - other (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Albumin, serum-low (hypoalbuminemia) (Metabolism and nutrition disorders) | 0 | 0 | 1 | 1 | 0 | 0
ALT, SGPT (serum glutamic pyruvic transaminase) (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0
AST, SGOT (serum glutamic oxaloacetic transaminase) (Metabolism and nutrition disorders) | 0 | 0 | 1 | 1 | 0 | 0
Bilirubin (hyperbilirubinemia) (Investigations) | 0 | 0 | 1 | 0 | 0 | 0
Creatinine (Investigations) | 0 | 1 | 0 | 0 | 0 | 0
GGT (gamma-glutamyl transpeptidase) (Investigations) | 0 | 0 | 1 | 0 | 0 | 0
Sodium, serum-low (hyponatremia) (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0
Confusion (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0
INR (International Normalized Ratio of Prothrombin time) (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Phase I: 36 Gy (N=3) | Phase I: 42 Gy (N=6) | Phase I: 40 Gy (N=5) | Phase I: 48 Gy (N=3) | Phase II Childs A (N=39) | Phase II Childs B (N=21)
Hemoglobin (Investigations) | 0 | 5 | 4 | 2 | 29 | 15
Leukocytes (total WBC) (Investigations) | 1 | 3 | 2 | 2 | 31 | 16
Neutrophils/Granulocytes (ANC/AGC) (Investigations) | 0 | 0 | 1 | 1 | 19 | 5
Platelets (Investigations) | 1 | 4 | 4 | 2 | 35 | 21
INR (international normalized ratio of prothrobin time) (Investigations) | 3 | 3 | 5 | 2 | 20 | 18
PTT (partial thromboplastin time) (Investigations) | 0 | 2 | 0 | 1 | 11 | 7
Ascites (non-malignant) (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Diarrhea (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Albumin, Serum-low(hypoalbuminemia) (Metabolism and nutrition disorders) | 2 | 6 | 5 | 1 | 30 | 21
Alkaline Phosphate (Metabolism and nutrition disorders) | 0 | 4 | 4 | 3 | 21 | 15
ALT, SGPT (Metabolism and nutrition disorders) | 2 | 1 | 3 | 2 | 29 | 14 — Serum Glutamic Pyruvic Transaminase
AST, SGOT (Metabolism and nutrition disorders) | 2 | 5 | 5 | 3 | 38 | 21 — Serum Glutamic oxaloacetic Transaminase
Bilirubin (Investigations) | 3 | 5 | 5 | 3 | 33 | 21 — Hyperbilirubinemia
Calcuim, Serum-Low (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0 — hypocalcemia
Creatinine (Investigations) | 0 | 0 | 2 | 0 | 12 | 4
GGT (Investigations) | 3 | 5 | 3 | 3 | 35 | 18 — Gamma-Glutamyl Transpeptidase
Potassium (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 — Serum high Hyperkalemia
Sodium (Metabolism and nutrition disorders) | 0 | 2 | 1 | 0 | 12 | 6 — Serum-low hypokalemia
Potassium (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 5 | 2 — Serum-Low- Hypokalemia
Muscle Weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 — Whole body- generalized
Pain (Gastrointestinal disorders) | 1 | 2 | 1 | 0 | 0 | 0 — Abdomen pain
Urinary frequency/urgency (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes